CLINICAL TRIAL: NCT04150380
Title: Biological Signature and Safety of an Immunomodulatory Probiotic Intervention for Veterans With PTSD
Brief Title: Probiotic (LGG) for Veterans With PTSD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Collaborators: University of Colorado, Denver (Other); University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Lisa Brenner, Director of the VHA Rocky Mountain MIRECC, VA Eastern Colorado Health Care System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-2415
Record Dates: First submitted 2019-10-18; First posted 2019-11-04 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Post Traumatic Stress Disorder; Inflammation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Inflammation

STUDY DESIGN:
Intervention Model Description: longitudinal, double blind, randomized placebo-controlled design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Supplement (Experimental): 8 weeks of dietary augmentation with oral LGG 1.0 x 1010 colony forming units (CFU) once daily (delivered in a size 1 capsule)
  Interventions: Biological: Lactobacillus rhamnosus GG (LGG; ATCC strain 53103; CRMTS #11272; PTS #3766)
- Placebo (Placebo Comparator): 8 weeks of dietary augmentation with placebo once daily (delivered in a size 1 capsule)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Lactobacillus rhamnosus GG (LGG; ATCC strain 53103; CRMTS #11272; PTS #3766) — See arm descriptions
  Arms: Supplement
Other: Placebo — See arm descriptions
  Arms: Placebo

SUMMARY:
Exaggerated inflammation in the body and brain is thought to play a role in the vulnerability to and aggravation and perpetuation of adverse consequences among those with posttraumatic stress disorder (PTSD). The proposed study begins the process of investigating the use of a natural immunoregulatory/anti-inflammatory probiotic, Lactobacillus rhamnosus GG (LGG; ATCC53103), to treat chronic symptoms associated with PTSD among Veterans. By looking at the impact of probiotic supplementation on biological signatures of increased inflammation, as reflected by biomarkers of inflammation, gut microbiota composition, intestinal permeability, stress response, decision making, and PTSD symptoms, this study may identify a novel intervention for the treatment of symptoms associated with this frequently occurring condition.

DETAILED DESCRIPTION:
United States military Veterans from recent conflicts are coping with symptoms related to posttraumatic stress disorder (PTSD). Many Veterans are resistant to conventional health and mental health interventions (e.g., medication, psychotherapy), and often symptoms are not significantly improved by traditional treatments. Alternative treatment methods are needed. An underlying feature of PTSD is exaggerated inflammation, both peripherally and in the central nervous system, which is thought to play an important role in the vulnerability to, aggravation of, and perpetuation of adverse consequences of this condition. Therefore, an innovative intervention strategy would be the use of immunoregulatory/anti-inflammatory probiotics to reduce inflammation. In this study, the investigators will investigate the effects of an 8-week oral administration of an immunoregulatory probiotic, Lactobacillus rhamnosus GG (LGG; ATCC53103), a probiotic shown to have anti-inflammatory and immunoregulatory effects (i.e., decreases in C-reactive protein [CRP]). Project aims will be assessed using a longitudinal, double blind, randomized placebo-controlled design. After initial evaluation procedures to confirm PTSD diagnosis, 59 participants will be randomized to probiotic supplementation and 59 will be randomized to placebo supplementation.

Primary Aim. Demonstrate the effects of LGG in a cohort of OEF/OIF Veterans with PTSD and Functional Bowel Disorders (FBD), including IBS, on plasma CRP concentrations (mechanistic, primary outcome), and PTSD symptom severity (clinical, exploratory). Additional biological signatures associated with this condition will be considered exploratory, including gut microbial community and intestinal permeability [IP]), other biological signatures of inflammation, as well as stress responsivity and decision making. Hypothesis 1.1. Those who receive LGG supplementation will respond with lower plasma levels of CRP as compared to those allocated to placebo. Exploratory Hypothesis 1.2. Those who receive LGG supplementation will respond with decreased PTSD symptoms (PCL-5), as compared to those allocated to placebo. Exploratory Hypothesis 1.3. Those who receive LGG supplementation will respond with increased abundance of LGG and community-level shifts (e.g.,increased alpha diversity) in the gut microbiota (measured using qRT-PCR and DNA sequencing of the 16S rRNA gene, respectively), decreases in IP (decreased fatty acid binding protein 215 and D-amino acid oxidase16), increases in plasma concentrations of anti-inflammatory biomarkers (IL-10, IL-4), decreases in additional plasma biomarkers of inflammation (IL-6, IL-8, IFNγ, IL- 1α, IL-1β, and IL-12p70), reduced stress response (biological and psychological) during and after Cyberball, and improved decision-making (measured by performance on the modified Iowa Gambling Test [mIGT]) as compared to those allocated to placebo. Exploratory Hypothesis 1.4. The effect of LGG supplementation on stress response, decision-making, and PTSD symptom severity is mediated by effects of LGG supplementation on the gut microbiota, intestinal permeability, and plasma biomarkers of inflammation.

ELIGIBILITY:
Inclusion criteria

* History of at least one deployment in support of OEF/OIF
* Current diagnosis of PTSD per the Clinician Administered PTSD Scale-5 (CAPS-5)
* Current diagnosis of Functional Bowel Disorder by ROME IV
* CRP level of 1.0 mg/L or above at baseline
* Medical clearance to participate by study providers
* Age between 18 and 60
* Ability to provide informed consent
* Willingness to abstain from probiotic supplements (pills, tablets, oils, foods, etc.) other than the investigational product provided until all study procedures are completed
* Willingness to provide blood and stool samples

Exclusion criteria

* Inability to adequately respond to questions regarding the informed consent procedure
* Currently involved in the criminal justice system as a prisoner or ward of the state
* Non-English speaking
* Current (past month) alcohol or substance abuse or dependence
* Lifetime history of bipolar disorder or psychosis or anxiety disorders (excluding PTSD).
* Consistent (e.g., 5x/week or greater) probiotic supplementation within the last month, including probiotic food products such as yogurt, as determined by phone screen interview and Probiotic Food Check List
* Receiving intravenous, intramuscular, or oral antibiotics within the last month
* Presence of central venous catheters (CVCs)
* Gastrointestinal (GI) barriers as identified by the 2-week run-in period as determined by the study team
* Participation in conflicting interventional research protocol
* Vital signs outside of acceptable range, i.e., blood pressure >160/100, pulse >100
* Use of any of the following drugs within the last 6 months: antifungals, antivirals or antiparasitics (intravenous, intramuscular, or oral); oral, intravenous, intramuscular, or inhaled corticosteroids; cytokines or cytokine inhibitors; methotrexate or immunosuppressive cytotoxic agents
* Acute disease at the time of enrollment (defer sampling until the participant recovers). Acute disease is defined as the presence of a moderate or severe illness with or without fever (e.g., oral temperature >100° F)
* Any medical condition deemed exclusionary by the Principal Investigators
* History of cancer
* Unstable dietary history as determined by the PIs (e.g., major changes in diet during the previous month, where the subject has eliminated or significantly increased a major food group in the diet)
* Positive test for human immunodeficiency virus (HIV), Hepatitis B virus, or Hepatitis C virus
* Any confirmed or suspected condition/state of immunosuppression or immunodeficiency (primary or acquired) including HIV infection, or those receiving immunosuppressive drugs or treatment including antineoplastic therapy, post-transplantation immunosuppressive therapy, and/or radiation therapy
* Major surgery of the GI tract, with the exception of cholecystectomy and appendectomy, in the past five years. Any major bowel resection at any time
* Female who is pregnant or lactating
* Treatment for or suspicion of ever having had toxic shock syndrome
* History of moderate and/or severe traumatic brain injury

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 383 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of C-reactive protein (CRP) | Change from basline to directly following the 8 week intervention
  Blood biomarker of inflammation

SECONDARY OUTCOMES:
PTSD symptoms per the PTSD Checklist for DSM-5 (PCL-5) | Change from basline to directly following the 8 week intervention
  PTSD symptoms
Type and abundance measurement of gut microbiota | Change from basline to directly following the 8 week intervention
  qRT-PCR and DNA sequencing of the 16S rRNA gene
Plasma concentration of intestinal permeability | Change from basline to directly following the 8 week intervention
  fatty acid binding protein 2 and D-amino acid oxidase
Plasma concentration of inflammatory markers | Change from basline to directly following the 8 week intervention
  IL-10, IL-4, IL-6, IL-8, IFNy, IL-1a, IL-1b, and IL-12p70
Biological and psychological stress response | Immediately post-intervention
  Cyberball
Decision-making | Immediately post-intervention
  Iowa Gambling Test

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Brenner, Ph.D., Principal Investigator — US Department of Veterans Affairs
Locations (1):
- VA Rocky Mountain Regional Center, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No